CLINICAL TRIAL: NCT00439439
Title: ACHAT-STUDY: Argon-Beamer-Ablation of Cervical Heterotopic Gastral Mucosa, an Alternative Treatment of Chronic Globus Sensations - "Sham-Controlled" Multicenter Study
Brief Title: ACHAT-STUDY, Alternative Treatment of Chronic Globus Sensations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: II: Medizinische Klinik, Technische Universität München
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1427/05
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Globus; Deglutition Disorders
MeSH Terms: conditions — Globus Sensation; Deglutition Disorders | interventions — Argon Plasma Coagulation

ARMS (2):
- A (Sham Comparator): Sham Procedure
  Interventions: Radiation: Beamer Ablation (Argon Plasma Coagulation)
- B (Active Comparator): Verum Beamer ablation of heterotopic gastric mucosa
  Interventions: Radiation: Beamer Ablation (Argon Plasma Coagulation)

INTERVENTIONS:
Radiation: Beamer Ablation (Argon Plasma Coagulation) — APC-Beamerablation of heterotopic gastric mucosa

SUMMARY:
Globus sensations are associated with gastroesophageal reflux disease as well as the presence of a gastric inlet patch. No controlled trial exists on whether ablation of the cervical heterotopic mucosa may lead to improvement of chronic globus sensations. The aim of this sham-controlled trial is to clarify whether argon-beamer-ablation of cervical heterotopic gastric inlet patches of the esophagus improves patients' chronic globus sensations.

DETAILED DESCRIPTION:
Some data suggest that ablation of gastric inlet patches by argon beamer therapy might lead to alleviation of chronic globus sensation or sore throat. Acid reflux or its treatment is unlikely to influence these results (Meining et al. Argon plasma ablation of gastric inlet patches in the cervical esophagus may alleviate globus sensation: a pilot trial. Endoscopy. 2006 Jun;38(6):566-70). Within the present study we will perform a randomized, sham-controlled and blinded trial, where patients with heterotopic gastric mucosa (HGM) of the cervical esophagus and globus sensations (a chronic or intermittent lump in the throat for at least 3 months) are going to be randomized after histological verification of HGM in the study center (Technical University Clinic Munich). Either a beamer ablation of HGM or a sham-therapy will be performed after patients complete a validated questionnaire. Patients are blinded for 3 months, then after completing another questionnaire endoscopy is repeated.

ELIGIBILITY:
Inclusion Criteria:

* Globus sensations and histologically verified heterotopic gastric mucosa of the cervical esophagus

Exclusion Criteria:

* Malignancy in the ear, nose, and throat (ENT)-field
* Scleroderma
* Mental disability affecting a patient's ability to sign an informed consent document

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
outcome verified by a questionnaire (I.J. Deary et al) before therapy and follow up after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, MD, Principal Investigator — II. Medical Department, TU-Munich
Locations (1):
- II. Medical Department, Technical University Munich, Munich, Bavaria, Germany

REFERENCES:
- [Background] Meining A, Bajbouj M, Preeg M, Reichenberger J, Kassem AM, Huber W, Brockmeyer SJ, Hannig C, Hofler H, Prinz C, Schmid RM. Argon plasma ablation of gastric inlet patches in the cervical esophagus may alleviate globus sensation: a pilot trial. Endoscopy. 2006 Jun;38(6):566-70. doi: 10.1055/s-2006-925362. PMID 16802267